CLINICAL TRIAL: NCT00824200
Title: Behavior and Exercise Versus Drug Treatment in Men With Nocturia
Brief Title: Behavior and Exercise Versus Drug Treatment in Men With Nocturia (BEDTiMe)
Acronym: BEDTiMe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Atlanta VA Medical Center (U.S. Federal Agency)
Collaborators: Emory University (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Theodore Johnson II, M.D., M.P.H., Site Director, Birmingham/Atlanta VA GRECC, Atlanta VA Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: VA RR&D No. D6110R; D6110R (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Nocturia
Keywords: Sleep; Quality of life; nocturia
MeSH Terms: conditions — Nocturia | interventions — Tamsulosin

STUDY DESIGN:
Intervention Model Description: Factorial design with no true placebo arm- drug alone versus behavior alone versus drug + behavior
Who Masked: Outcomes Assessor
Masking Description: Main outcome measure was 7-day bladder diary derived count of nocturia episodes. Assessor was blinded to randomization
Oversight: Data Monitoring Committee: No

ARMS (3):
- Behavioral and Exercise Therapy (M-BET) (Experimental): Multicomponent behavior and exercise therapy program (M-BET) - pelvic floor muscle exercises, urge suppression strategies, fluid strategies, sleep hygiene & non-pharmacological management of peripheral edema. M-BET alone will be given with placebo capsules.
  Interventions: Behavioral: Behavioral; Drug: placebo
- Drug Therapy w/ Behavioral Placebo (Active Comparator): alpha-adrenergic antagonist medication with a placebo behavioral intervention
  Interventions: Drug: tamsulosin (alpha-adrenergic antagonist medication); Behavioral: placebo
- Combination Therapy (Active Comparator): Combination therapy: MBET and alpha-adrenergic antagonist medication
  Interventions: Behavioral: Behavioral; Drug: tamsulosin (alpha-adrenergic antagonist medication)

INTERVENTIONS:
Behavioral: Behavioral — Multicomponent Behavioral and Exercise Therapy (M-BET) - pelvic floor muscle exercises, urge suppression strategies, fluid strategies, sleep hygiene & non-pharmacological management of peripheral edema.
  Other Names: M-BET
  Arms: Behavioral and Exercise Therapy (M-BET); Combination Therapy
Drug: tamsulosin (alpha-adrenergic antagonist medication) — 0.4 mg given daily
  Other Names: Drug Group
  Arms: Combination Therapy; Drug Therapy w/ Behavioral Placebo
Drug: placebo — tamsulosin placebo
  Arms: Behavioral and Exercise Therapy (M-BET)
Behavioral: placebo — placebo behavioral intervention
  Other Names: Face Recognition Behavioral placebo
  Arms: Drug Therapy w/ Behavioral Placebo

SUMMARY:
Nocturia, waking at night from sleep to void, is a prevalent and troublesome symptom. Treatment with an alpha-adrenergic antagonist medication (α-blockers) is a standard therapy for LUTS in men, but α-blockers offer only limited reductions in nocturia. While combinations of multiple drugs could be used, many individuals wish to take fewer medications.

Participants in the BEDTiMe Nocturia Study will undergo a series of visits during which they will receive a combination of either standard drug therapy (or placebo) and a behavioral intervention tailored to help with nocturia or problems with nocturia. Participants will be evaluated for outcomes at 12 weeks and followed for six months.

This study will yield important information related to alternative treatments of nocturia in men, as well as novel information regarding the clinical importance of these nocturia reductions. This study has the potential to alter standards of care.

DETAILED DESCRIPTION:
Nocturia, waking at night from sleep to void, is a prevalent and troublesome symptom. While other lower urinary tract symptoms (LUTS)-- including poor urinary stream, urgency, frequency, and straining to void-- are also common, nocturia is one of the most bothersome LUTS. Nocturia causes sleep disruption and is associated with accidental falls and higher utilization of sick days from work. Conditions that result in low volume urinary voids, high urine production at night, and/or primary sleep disturbances will cause nocturia. Overactive bladder (OAB), benign prostatic hyperplasia (BPH), congestive heart failure (CHF), poorly controlled diabetes mellitus (DM), peripheral edema, and obstructive sleep apnea all cause nocturia. Individual patients frequently have multiple conditions potentially related to nocturia, which highlights the need for strategies that are broad-based interventions. Treatment with an alpha-adrenergic antagonist medication (α-blockers) is a standard therapy for LUTS in men, but α-blockers offer only limited reductions in nocturia. While combinations of multiple drugs could also be employed to more successfully treat nocturia, non-drug treatments are an important option for those unwilling or unable to take additional medications.

The BEDTiMe Nocturia Study (Behavior and Exercise or Drug Trial in Men with Nocturia), is a two-site (Atlanta and Birmingham), randomized, clinical trial. The 200 male participants will be stratified by degree of nocturia and urinary flow rate and randomized to three treatment arms: 1) α-blocker therapy alone; versus 2) a standardized, multicomponent behavioral and exercise therapy (M-BET), given with placebo tablets; versus 3) combination therapy (M-BET and α-blockers). The M-BET intervention includes: training in pelvic floor muscle rehabilitation, self monitoring with bladder diaries, and teaching urge suppression and other skills to inhibit detrusor contractions; fluid management strategies; sleep hygiene strategies; and non-pharmacological management of lower extremity edema. Interventions similar to M-BET have shown reductions in nocturia in women with urge urinary incontinence (UI) that exceeded benefit from anticholinergic drug therapy. The use of this intervention in men builds upon strong pilot data from the MINIM trial (Multicomponent Interventions for Nocturia in Men; VA GRECC Pilot, VA Medical Research Services) and the ongoing study Behavioral Treatment For Overactive Bladder In Men (VA RR&D B02-2489R, Burgio, PI).

The study design allows 3 main research questions to be addressed: 1) Does M-BET reduce nocturia more than α-blockers?; 2) Does M-BET improve sleep more than α-blockers?; and 3) Will combination therapy be more effective than either treatment alone? The main outcomes will be nocturia reduction and sleep improvement at 12 weeks. Nocturia reduction will be assessed by participant completed bladder diaries and sleep improvement will be assessed by wrist-actigraph determined sleep efficiency, total sleep time, and wake time after sleep onset.

This study will yield important information related to alternative treatments of nocturia in male veterans, as well as novel information regarding the clinical importance of these nocturia reductions. Though many clinicians employ single-agent α-blockers routinely for the treatment of nocturia, few utilize multicomponent behavioral interventions or use behavioral therapy. Thus, this study has the potential to alter standards of care.

ELIGIBILITY:
Inclusion Criteria:

1. Nocturia ≥2 episodes / night average on the screening diary;
2. Willingness and appropriateness to receive an α- blocker;
3. Willingness to keep a bladder and sleep diary;
4. Willingness to wear a wrist actigraph; and
5. Willingness to make study visits

Exclusion Criteria:

1. Evidence of overt bladder outlet obstruction: peak uroflow <4 mL/sec on a void of ≥125 mL, or a PVR of ≥ 300 mL;
2. Use of clean intermittent self-catheterization at home or having been instructed by a provider to do so within the last 12 months;
3. Genitourinary cancer, including active prostate cancer with ongoing surgical or radiation treatment, or the need of treatment, or bladder cancer, or persistent unexplained hematuria;
4. Obstructive sleep apnea with CPAP use, provider diagnosis with symptoms, or strong suspicion of diagnosis during screening;
5. Having Parkinson's disease with an uncontrolled tremor (invalidates wrist actigraphy);
6. Poorly controlled congestive heart failure as evidenced on physical examination;
7. Poorly controlled diabetes mellitus with either hemoglobin A1c of ≥ 7.5 or a random glucose ≥ 200 within last 3 months; or
8. Unstable health conditions expected to result in death or hospitalization within 3 months, as assessed by PI or Site PI;
9. Previously receiving intensive bladder training;
10. Allergic to Tamsulosin;
11. Previous spinal cord injury;
12. Currently on dialysis or in consideration for dialysis due to end stage renal disease;
13. More than 2 urinary tract infections within the last 12 months;
14. Not able to transfer independently from a wheelchair to the toilet;
15. Unstable dose of diuretic within the past 3 months;
16. Has an artificial urinary sphincter;
17. Impaired mental status;
18. TURP or other urologic surgery within the last 6 months.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-07; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Nocturia episodes (voiding diary) | 12 weeks
  Participant recorded bladder diary over 7-day that included nocturia episodes

SECONDARY OUTCOMES:
Sleep quality | 12 weeks
  Pittsburgh Sleep Quality Index
Bother from nocturia | 12 weeks
  American Urological Association 7 symptom index accompanying bother index; specific question on nocturia
Symptom-specific quality of life measure | 12 weeks
  The International Consultation on Incontinence Nocturia Quality of Life Instrument (ICI-NQOL)
Nocturia episodes (self report) | 12 weeks
  The 7th question on the American Urological Association 7 Symptom Index: "Over the past month, how many times did you most typically get up to urinate from the time that you went to bed at night until the time you got up in the morning? 0, 1, 2, 3, 4 or 5 or more.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Johnson II, MD, MPH, Principal Investigator — Atlanta Veteran Affairs Adminstration, Emory University School of Medicine
Locations (2):
- United States (2):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - Atlanta VA Medical Center, Atlanta, Georgia

REFERENCES:
- [Result] Johnson TM 2nd, Vaughan CP, Goode PS, Bliwise DL, Markland AD, Huisingh C, Redden DT, McGwin G, Eisenstein R, Ouslander JG, Issa M, Burgio KL. Pilot Results from a Randomized Trial in Men Comparing Alpha-Adrenergic Antagonist versus Behavior and Exercise for Nocturia and Sleep. Clin Ther. 2016 Oct 28:S0149-2918(16)30742-1. doi: 10.1016/j.clinthera.2016.10.001. Online ahead of print. PMID 28029383